CLINICAL TRIAL: NCT04772092
Title: Impact of Age and Geriatric Co-morbidities on Lymphocyte Phenotype in Patients 70 Years of Age and Older
Acronym: PHENOGERIA
Status: Withdrawn | Type: Observational
Why Stopped: Departure from the department of the principal investigator
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BARBEN 2020
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Geriatrics Immunosenescence
MeSH Terms: interventions — Blood Specimen Collection; Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Seniors: 70 years of age and over, inpatients or outpatients
  Interventions: Biological: Blood samples; Other: Data collection

INTERVENTIONS:
Biological: Blood samples — during the routine blood test, collection of additional blood samples:
  * 1 x 5 mL heparinized tube for plasma collection and storage
  * 1 heparinized 5 mL tube for immunophenotyping
  * 4 x 10 mL EDTA tubes for white blood cell (WBC) collection and cryopreservation
Other: Data collection — * clinical examination data
  * test results to measure the degree of geriatric fatigability
  * Frailty screening questionnaire for neoplasia patients (G8 score)

SUMMARY:
An individual's immune profile changes with age, and can sometimes be involved in the development of certain diseases such as infections or cancers, in a process called immunosenescence. Some data tend to show that there is a link between this immune profile and geriatric fragility (autonomy, difficulties with walking, memory, undernutrition, co-morbidities, depression). The aim of this study is to describe this profile, or immune phenotype, and to see if there is a link with the different aspects of geriatric assessment in patients without cancer or infection. In addition, these data will serve as a basis for comparison with the same analyses performed on breast cancer patients at the Centre Georges François Leclerc.

ELIGIBILITY:
Inclusion Criteria:

* Person who has not opposed to inclusion in the study
* Male or female aged 70 and over admitted to the Champmaillot Geriatric Center on an inpatient or outpatient basis.

Exclusion Criteria:

* Person not affiliated to national health insurance system
* Person subject to a measure of legal safeguard (curatorship, etc)
* Person with an acute infection
* Person with suspected cancer or active cancer
* Long-term immunosuppressive or corticosteroid therapy
* HIV and/or HBV and/or HCV positive serology

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: A person at least 70 years of age admitted to the Champmaillot Geriatric Center on an inpatient or outpatient basis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
percentage of immune cells in peripheral blood | At inclusion
  technique used: flow cytometry